CLINICAL TRIAL: NCT02776280
Title: Oral Fluoride Bioavailability by the Consumption of Meals Prepared With Fluoridated Water or Salt
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Livia Maria Andaló Tenuta, Associate Professor, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: FOPBioq006
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Fluoridation
Keywords: water; salt; oral fluids; plaque; dental caries
MeSH Terms: conditions — Plaque, Amyloid; Dental Caries | interventions — Meals

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Negative control (Placebo Comparator): Meal prepared with non-fluoridated water and salt
  Interventions: Other: Meal
- Fluoridated water (Experimental): Meal prepared with fluoridated water
  Interventions: Other: Meal
- Fluoridated salt (Experimental): Meal prepared with fluoridated salt
  Interventions: Other: Meal

INTERVENTIONS:
Other: Meal — Typical Brazilian meal consisting of rice, beans and meat with vegetables

SUMMARY:
This study will assess the concentration of fluoride in saliva and dental biofilm (fluid and solids) during and up to 2 hours after the consumption of typical Brazilian meals prepared with fluoridated water (0.7 ppm F) or fluoridated salt (250 mg F/kg). Typical Brazilian meals (rice, beans, meat with vegetables) will be prepared using fluoridated water, salt, or non-fluoridated water and salt. In an crossover design, twelve volunteers will eat 4.67 g of food/kg body weight of each meal, on fasting, during 15 min. Before the ingestion, unstimulated saliva and dental biofilm will be collected for determination of fluoride concentration. During the meal, 3 samples of the alimentary bolus (at 5, 10 and 15 min of mastication) will be collected for determination of fluoride concentration. Dental biofilm will be collected immediately after the ingestion of the meal. Saliva will then be collected after 5, 10, 15, 30, 60 and 120 min. All samples will be analyzed for fluoride using an ion-specific electrode. In order to standardize biofilm formation, during lead-in and wash-out periods, volunteers will: 1. brush their teeth with non-fluoride toothpaste; 2. refrain from brushing superior posterior teeth for 2 days before each phase; and 3. chew sucrose-containing chewing gum 5 times/day, for 10 min, during the 2 days prior to each phase. Groups will be compared by ANOVA and Tukey test.

ELIGIBILITY:
Inclusion Criteria:

* good general health
* good oral health
* not having used topical fluorides in the last 2 months

Exclusion Criteria:

* poor general health
* poor oral health
* breastfeeding
* expecting mothers

Ages: 18 Years to 33 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Fluoride concentration in the alimentary bolus | up to 15 min after start of the meal
Fluoride concentration in saliva | up to 120 min after meal
Fluoride concentration in dental biofilm | up to 120 min after the meal

IPD SHARING:
Plan to Share IPD: No